CLINICAL TRIAL: NCT00058006
Title: Pilot Randomized Trial Of Adjuvant Celecoxib In Patients With Early Stage Head And Neck And Non-Small Cell Lung Cancers
Brief Title: Celecoxib in Treating Patients With Early-Stage Head and Neck Cancer or Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: NU 02V2; NU-02V2; PHARMACIA-NU-02V2
Record Dates: First submitted 2003-04-07; First posted 2003-04-09 (Estimated); Last update posted 2012-06-11 (Estimated); Status verified 2012-06

CONDITIONS: Head and Neck Cancer; Lung Cancer
Keywords: stage I non-small cell lung cancer; stage I squamous cell carcinoma of the hypopharynx; stage I squamous cell carcinoma of the larynx; stage I squamous cell carcinoma of the lip and oral cavity; stage I squamous cell carcinoma of the nasopharynx; stage I squamous cell carcinoma of the oropharynx; stage I squamous cell carcinoma of the paranasal sinus and nasal cavity; stage II squamous cell carcinoma of the hypopharynx; stage II squamous cell carcinoma of the larynx; stage II squamous cell carcinoma of the lip and oral cavity; stage II squamous cell carcinoma of the nasopharynx; stage II squamous cell carcinoma of the oropharynx; stage II squamous cell carcinoma of the paranasal sinus and nasal cavity; salivary gland squamous cell carcinoma; stage I salivary gland cancer; stage II salivary gland cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Squamous Cell Carcinoma of Head and Neck; Salivary Gland Neoplasms | interventions — Celecoxib; Chemotherapy, Adjuvant

INTERVENTIONS:
Drug: celecoxib
Procedure: adjuvant therapy

SUMMARY:
RATIONALE: Chemoprevention therapy is the use of certain drugs to try to prevent the development or recurrence of cancer. The use of celecoxib may be an effective way to prevent the recurrence of stage I or stage II head and neck cancer or stage I non-small cell lung cancer.

PURPOSE: This randomized phase II trial is studying celecoxib to see how well it works compared to that of a placebo in preventing disease recurrence in patients with stage I or stage II head and neck cancer or stage I non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the rate of new malignancies (recurrences and second primary tumors) in patients with early-stage head and neck cancer or non-small cell lung cancer treated with celecoxib vs placebo.
* Compare the event-free and overall survival of patients treated with this drug vs placebo.
* Determine the toxic effects associated with long-term use of celecoxib in these patients.
* Correlate cyclooxygenase-2 and transforming growth factor (TGF)-beta expression and CYP2C9 and TGF-beta genotypes with the rate of new malignancies and survival of patients treated with this drug vs placebo.

OUTLINE: This is a randomized, placebo-controlled, double-blind, multicenter study. Patients are stratified according to smoking history (active smokers [including those who quit within 1 year of diagnosis] vs former smokers vs non-smokers), tumor type (lung cancer vs head and neck cancer), and stage (I vs II for head and neck cancer or T1 vs T2 for lung cancer). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral celecoxib twice daily.
* Arm II: Patients receive oral placebo twice daily. In both arms, treatment continues for 24 months in the absence of disease recurrence or unacceptable toxicity.

Patients are followed every 6 months for 5 years or until disease recurrence.

PROJECTED ACCRUAL: A total of 121 patients (approximately 60 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* One of the following histologically confirmed diagnoses:

  * Stage I non-small cell lung cancer (NSCLC)

    * No small cell component
  * Stage I-II squamous cell cancer of the head and neck

    * No WHO type II or III nasopharyngeal cancer
    * No sinonasal undifferentiated carcinoma
* No evidence of disease
* Must have undergone surgery or radiotherapy with curative intent within the past 4-24 weeks

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-1

Life expectancy

* Not specified

Hematopoietic

* Platelet count at least 50,000/mm^3

Hepatic

* Bilirubin normal
* AST/ALT no greater than 2 times upper limit of normal

Renal

* Creatinine no greater than 2.0 mg/dL

Cardiovascular

* No uncontrolled hypertension
* No severe congestive heart failure

Pulmonary

* No history of asthma caused by cyclooxygenase-2 (COX-2) inhibitors, nonsteroidal anti-inflammatory drugs (NSAIDs), salicylates, or sulfonamides

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after study participation
* No other prior malignancy (including skin cancer and in situ malignancies)
* No diagnosis of peptic ulcer disease or gastritis/esophagitis within the past 60 days
* No prior hypersensitivity reaction to COX-2 inhibitors, NSAIDs, salicylates, or sulfonamides
* No other concurrent medical condition that would preclude study compliance

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* No cumulative oral or IV corticosteroid use totalling more than 2 weeks within the past 3 months
* No concurrent oral steroids for more than 2 consecutive weeks
* Concurrent inhaled steroids allowed

Radiotherapy

* See Disease Characteristics
* No prior definitive radiotherapy for stage I NSCLC

Surgery

* See Disease Characteristics
* Prior pneumonectomy or lobectomy with mediastinal lymph node sampling or dissection for stage I NSCLC allowed
* No prior segmentectomies or wedge resections for stage I NSCLC

Other

* More than 60 days since prior treatment for peptic ulcer disease or gastritis/esophagitis
* No prior NSAID use within the past 30 days at a frequency of 3 or more times a week for more than 2 weeks
* No concurrent NSAIDs (including low-dose aspirin)
* No other concurrent COX-2 inhibitors
* No concurrent fluconazole
* No concurrent lithium

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-09; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Athanassios Argiris, MD, Study Chair — Robert H. Lurie Cancer Center
Locations (4):
- United States (4):
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - Rush Cancer Institute at Rush University Medical Center, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina